CLINICAL TRIAL: NCT03842995
Title: South-seq: DNA Sequencing for Newborn Nurseries in the South
Brief Title: South-seq: Deoxyribonucleic Acid (DNA) Sequencing for Newborn Nurseries in the South
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Mississippi Medical Center (Other); HudsonAlpha Institute for Biotechnology (Other); Woman's Hospital, Louisiana (Other); Children's Hospital New Orleans, LA (Other); Norton's Children's Hospital (Unknown); University of Louisville (Other)
Responsible Party: Principal Investigator, Maria Danila, MD, MSc, MSPH, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300000328; U01HG007301 (NIH)
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Whole Genome Sequencing
Keywords: Genetic Counseling; NICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetic Counselor (Placebo Comparator): Standard of Care. Parents/caregivers of neonates enrolled in SouthSeq will receive counseling on their child's Whole Genome Sequencing (WGS) results from Genetic Counselors
  Interventions: Behavioral: Genetic Counselor
- Trained Healthcare Provider (Experimental): Healthcare providers (e.g., neonatologists and neonatology nurse practitioners) will receive training to competently deliver Whole Genome Sequencing results to parents/caregivers of neonates enrolled in SouthSeq
  Interventions: Behavioral: Trained Healthcare Provider

INTERVENTIONS:
Behavioral: Genetic Counselor — Standard of Care
  Arms: Genetic Counselor
Behavioral: Trained Healthcare Provider — Neonatologists and Neonatology Nurse Practitioners that receive training to deliver whole genome sequencing results
  Arms: Trained Healthcare Provider

SUMMARY:
2,000 infants with signs suggestive of a genetic disorder being treated at a neonatal intensive care unit (NICU) in which African-American and rural populations are highly represented will be enrolled. Whole genome sequencing (WGS) will be used to identify pathogenic variation in DNA from these infants. Stakeholders, including parents, clinicians, and community leaders, will be engaged to develop culturally adapted educational materials and to equip non-genetics providers to return WGS results. Parents will be provided with these materials through a web portal, the Genome Gateway, and will be placed into one of two arms of a randomized trial to compare the effectiveness technology-assisted WGS result delivery by non-genetics providers relative to result delivery from genetic counselors.

DETAILED DESCRIPTION:
Barriers to widespread and routine implementation of WGS-enabled clinical care exist at several levels. Surveys of clinicians indicate discomfort in their understanding of genomics and ability to communicate results to patients, and also concern about the time required to do so. Medical geneticists and genetic counselors are disproportionately concentrated in large academic centers, and their numbers are inadequate to support the number of patients that may benefit from WGS. This limitation will have a disproportionate effect on patients in rural and/or medically underserved areas. For example, all but one of the genetic counselors in Alabama are based in Birmingham or Huntsville (lone exception is in Mobile), which means that the southern 2/3 of the state, including major rural underserved areas, have little to no local access to genetic counseling services.

These barriers are especially apparent in neonatal care. For parents of sick neonates, their first interactions with the healthcare system take place in the NICU. Neonatology training traditionally emphasizes critical care and can neglect communication, with one study reporting that 93% of fellows stated that their training in this area should be improved. There is a particular lack of training in genomic neonatal medicine, with few didactic lectures, role play sessions, simulated experiences, or hands on training in clinically relevant scenarios. When infants are diagnosed with congenital anomalies in utero, prenatal consultation with subspecialists can be confusing for genetic conditions with a spectrum of causes and outcomes, and inconsistent information given by different providers, e.g., the neonatologist and the pediatric surgeon.

A central premise underlying the proposal is that non-genetics health care providers, including those outside of academic medical centers, can be empowered to use WGS-testing in their practices. There is ample precedent for implementation of complex technology in primary care: pediatricians, internists, and family practitioners routinely use advanced imaging technologies without a deep understanding of the underlying technology. Bringing WGS-enabled genomic medicine to community health care providers requires, at the least, straightforward criteria to identify patients who may benefit, a user-friendly consent process, clearly worded laboratory reports, easily accessible patient education materials, ready access to support from medical geneticists and genetic counselors, and basic training in how WGS can be applied routinely. The study investigators seek to demonstrate that, if these factors are provided, WGS can be carried out and relevant results returned by newborn medicine providers, and that the patient experience will be at least equal to that achieved with the traditional approach of face-to-face counseling by a geneticist or genetic counselor.

In order to compare technology-assisted WGS result delivery by trained healthcare providers to formal genetic counseling by genetic counselors (standard of care), a series of surveys have been developed and will be completed online using the Genome Gateway platform/website developed for this trial. The survey time points are enrollment (specimen collection from the infant/proband), return of results (ROR) (roughly 2-3 months post-enrollment when WGS results are available), 1-month post-ROR counselling, 4-months post-ROR counselling, and 4.5 months post-ROR counselling.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregiver/guardian of a newborn (proband) who meets the inclusion criteria in Specific Aim 1
* Parent or caregiver/guardian is willing to participate and answer surveys

Exclusion Criteria:

* Proband has secondary findings from WGS
* Parent or caregiver is not available to participate and answer surveys
* Parent or caregiver requires language interpreter services/translated materials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Danila, MD, MSc,MSPH, Study Director — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham/Children's of Alabama, Birmingham, Alabama
  - Woman's Hospital, Baton Rouge, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biesecker BB, Woolford SW, Klein WMP, Brothers KB, Umstead KL, Lewis KL, Biesecker LG, Han PKJ. PUGS: A novel scale to assess perceptions of uncertainties in genome sequencing. Clin Genet. 2017 Aug;92(2):172-179. doi: 10.1111/cge.12949. Epub 2017 Jan 30. PMID 27925165
- [Background] Costal Tirado A, McDermott AM, Thomas C, Ferrick D, Harris J, Edwards A, McAllister M. Using Patient-Reported Outcome Measures for Quality Improvement in Clinical Genetics: an Exploratory Study. J Genet Couns. 2017 Oct;26(5):1017-1028. doi: 10.1007/s10897-017-0079-6. Epub 2017 Mar 9. PMID 28281044

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this clinical trial the participants were parents of neonates that had whole genome sequencing performed. Only the answers from mothers were analyzed, thus in this RCT only the mothers were enrolled/analyzed. Neither the neonates or the health-care providers were enrolled in this RCT. This was not a dyad study.
Period: Overall Study
Arm/Group | Genetic Counselor | Trained Healthcare Provider
Started | 240 | 237
Completed | 98 | 95
Not Completed | 142 | 142

BASELINE CHARACTERISTICS:
Population: There were 240 participants (i.e. mothers) in the genetic counselor group and 237 participants (i.e. mothers) in the trained healthcare provider group. This was not a dyad study. The neonates or healthcare providers were not enrolled as participants in this study. Only mothers participated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Genetic Counselor | Trained Healthcare Provider | Total
Number analyzed (Participants) | 240 | 237 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] — This was age of mother
  years | 27.29 (5.60) | 28.37 (5.84) | 27.82 (5.74)
Sex: Female, Male [Count of Participants; unit: Participants] — This study collected data on the mother of the child who had genome sequencing
  Participants
    Female | 240 | 237 | 477
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — This study collected race of mother
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 3 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 52 | 49 | 101
    White | 91 | 90 | 181
    More than one race | 7 | 7 | 14
    Unknown or Not Reported | 89 | 88 | 177

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Parental Empowerment Using the Genetic Counseling Outcome Scale (GCOS)
Description: Collected after return of whole genome sequencing results using the GCOS. The GCOS is a 24-item counseling outcome scale to assess parental empowerment through questions addressing five constructs: Decision control, Cognitive control, Behavioral control, Emotional regulation, and Future orientation. Each of the 24-items is answered with a 7-point Likert-type scale: Strongly disagree (1), Disagree (2), Slightly disagree (3), Neither agree nor disagree (4), slightly agree (5), agree (6), and strongly agree (7). Range of possible scores for those completing all items: 24-168. Higher scores are better.
Time Frame: 3 months post specimen collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetic Counselor | Trained Healthcare Provider
Number analyzed (Participants) | 98 | 95
score on a scale | 117.94 (13.85) | 117.19 (14.86)

2. Secondary Outcome: Evaluate Parental Uncertainties Using the Parental Perceptions of Uncertainties in Genomic Sequencing (PUGS)
Description: Collected after return of whole genome sequencing results using the PUGS. PUGS is an 8-item scale to assess uncertainties within three domains: Clinical, Affective, and Evaluative. Each of the questions is answered on a 5-point Likert-type scale: Very uncertain (1) to very certain (5). Range of possible scores for those completing all items: 8-40. Higher scores represent more certainty.
Time Frame: 3 months post specimen collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetic Counselor | Trained Healthcare Provider
Number analyzed (Participants) | 99 | 100
score on a scale | 29.11 (7.31) | 29.74 (5.87)

3. Secondary Outcome: Evaluate Personal Utility Using the Parental Personal Utility Scale (PrU)
Description: Collected after return of whole genome sequencing results using the PrU. This measure consists of 17 items answered with a 7-point Likert-type scale: Not at all useful (1), A little useful (2), Somewhat useful (3), Neutral (4), Useful (5), Very useful (6), and Extremely useful (7). Range of possible scores for those completing all items: 17-119. Higher scores are better.
Time Frame: 3 months post specimen collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genetic Counselor | Trained Healthcare Provider
Number analyzed (Participants) | 98 | 100
score on a scale | 78.40 (20.51) | 73.93 (19.86)

ADVERSE EVENTS:
Time Frame: Since the intervention in this study involved an educational intervention (healthcare providers were trained to deliver genetic results) no data on Adverse Events was collected.
Description: We did not collect data on mortality, or severe adverse events (e.g. hospitalization) in this study.
Arm/Group | Genetic Counselor | Trained Healthcare Provider
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This clinical trial did not include measures of mortality or adverse events. As safety reporting we counted the number of errors the trained healthcare providers made when delivering the genetic results to the parents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03842995/Prot_SAP_ICF_000.pdf